CLINICAL TRIAL: NCT06887621
Title: Patients at High Risk for Postoperative Nausea and Vomiting Undergoing Gynecological Surgery: Efficacy of Oral Amisulpride in Combination With Intravenous Ondansetron and Dexamethasone - a Parallel-group Randomized Trial
Brief Title: Efficacy of Adding Oral Amisulpride to Dual Prophylaxis for Postoperative Nausea and Vomiting in Patients at High Risk for Nausea and Vomiting Undergoing Gynecological Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, amsousa, MD, MsC, PhD, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 83804424.3.0000.0083
Record Dates: First submitted 2025-03-16; First posted 2025-03-20 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Nausea and Vomiting (PONV)
Keywords: Amisulpride; Postoperative Nausea and Vomiting; Laparoscopy; Gynecologic Surgical Procedures
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting | interventions — Color; Weights and Measures; Smell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo ● Dexamethasone 10 mg IV immediately after anesthesia induction ● Ondansetron 4 mg IV at the end of the surgical procedure.
  Interventions: Drug: Encapsulated placebo (matched for color, weight, smell and size)
- Oral Amisulpride (Experimental): Amisulpride 50 mg ● Dexamethasone 10 mg IV immediately after anesthesia induction ● Ondansetron 4 mg IV at the end of the surgical procedure.
  Interventions: Drug: Encapsulated amisulpride 50 mg (matched for color, weight, smell and size)

INTERVENTIONS:
Drug: Encapsulated amisulpride 50 mg (matched for color, weight, smell and size) — Amisulpride will be delivered orally 1 hour before anesthesia induction.
  Arms: Oral Amisulpride
Drug: Encapsulated placebo (matched for color, weight, smell and size) — Placebo will be delivered orally 1 hour before anesthesia induction.
  Arms: Placebo

SUMMARY:
Amisulpride is a potent antagonist of dopamine D2 and D3 receptors, both implicated in the emetic response when activated. It is currently used intravenously for the prevention of chemotherapy-induced and postoperative nausea and vomiting (PONV), but this route has a short half-life time of 4 to 5 hours, could be expensive, causes infusion-related pain, and is not available in Brazil. Some of these limitations could be overcome by the preemptive use of an oral formulation. At present, there are no data regarding the use of oral amisulpride for PONV, which is an affordable and painless option with half-life time of 12 hours. We propose a quadruple-blind clinical trial involving patients undergoing gynecological surgery aged 18 years and older, and assessed as being at high risk for PONV according to the Apfel Score (score 3 or 4). The primary outcome of this study is to evaluate complete response to PONV up to 24h, comparing the efficacy of adding 50 mg oral amisulpride as a third antiemetic agent to the standard institutional protocol at the Hospital da Mulher of São Paulo (IV dexamethasone 10 mg + IV ondansetron 4 mg) for laparoscopic surgeries. Secondary outcomes will evaluate (1) nausea, (2) vomiting, (3) nausea and vomiting, (4) use of rescue treatment, (5) overall adverse events, and (6) adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic hysterectomy to treat benign conditions.
* High risk for PONV according to the Apfel Score: scores 3 or 4.
* American Society of Anesthesiology (ASA) physical status: 1 or 2.

Exclusion Criteria:

* Cognitive or psychiatric conditions impairing consent or compliance.
* Incapability of using the mobile app MyCapp for data collection.
* History of allergy or sensibility to any medication included in the protocol: amisulpride, dexamethasone, ondansetron, fentanyl, midazolam, bupivacaine, morphine, propofol, rocuronium, sevoflurane, ephedrine, metaraminol, remifentanil, metamizole, ketoprofen, sugammadex, dimenhydrinate, pyridoxine hydrochloride, tramadol, dimethicone.
* Inability to swallow medications.
* Current use of typical or atypical antipsychotic medications.
* Gestation or lactation.
* Clinically significant cardiac arrhythmia or long QT syndrome documented.
* Hypokalemia (K+ < 3.5 mmol/L)
* Prolactin-dependent tumors.
* Pheochromocytoma.
* Parkinson's disease.
* Nausea or vomiting in the 24 hours before surgery.
* Therapeutic use of antiemetics, including corticosteroids.
* Emetogenic oncological therapy (above 10% probability of causing vomiting) in the 2 weeks before surgery.
* Persistent pre-operative hypotension on the day of surgery, defined as systolic blood pressure < 100 mmHg on at least 2 consecutive measurements.
* Mechanical ventilation plan or need for a naso/orogastric tube after surgery.
* Intestinal endometriosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-03-29 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with complete response | 24 hours after the end of anesthesia
  Complete response defined as the absence of emetic episodes (nausea, vomiting or retching) and no use of antiemetic medications.

SECONDARY OUTCOMES:
Time to first violation of the criteria for complete response | 24 hours after the end of anesthesia
  Time in minutes from the end of anesthesia until violation of criteria for complete response, defined as the absence of emetic episodes (nausea, vomiting or retching) and no use of antiemetic medications.
Number of participants with any nausea | 24 hours after the end of anesthesia
  Nausea (defined as unpleasant, subjective abdominal discomfort associated with the desire to vomit) measured on a 0 to 10 verbal response scale, in which 0 = no nausea at all and 10 = the worst nausea imaginable. "Any nausea" means a score ≥ 1.
Number of participants with vomiting | 24 hours after the end of anesthesia
  Any vomiting (expulsion of gastric contents) or dry-retching.
Number of participants with nausea and vomiting | 24 hours after the end of anesthesia
  Any nausea, vomiting, or dry-retching.
PONV Intensity | 24 hours after the end of anesthesia
  0 to 10 scale
Number of Participants Receiving Rescue Medication | 24 hours after the end of anesthesia
  Rescue medication defined as an antiemetic (or other medication) given with the intention of relieving nausea and/or vomiting and/or dry-retching, or any incidental use of a drug known to have antiemetic potential
Total number of adverse events | 48 hours after ingestion of the capsule
  Any adverse event
Number of serious adverse event | 48 hours after ingestion of the capsule
  Any adverse event classified as severe or life-threatening

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Sousa, MD, MsC, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital da Mulher, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers. Data shared will be coded, with no PHI included.
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).